CLINICAL TRIAL: NCT04870749
Title: Diagnostic Role of Visual Prostate Symptom Score and Intravesical Prostatic Protrusion in Male Lower Urinary Tract Symptoms
Brief Title: The Importance of Non-invasive Methods in the Diagnosis of Lower Urinary System Symptoms.
Status: Completed | Type: Observational
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Huseyin Saygin, Assistant Professor Department of Urology, Cumhuriyet University
Other Study IDs: CumhuriyetU urology
Record Dates: First submitted 2021-04-27; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Urinary Obstruction
Keywords: IPP; IPSS; VPSS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- lower urinart tract syptoms: Lower urinary tract symptoms (LUTS) are common in older men and one of the main reasons for this is the enlargement in prostate gland volume caused by hormonal changes.
  Interventions: Diagnostic Test: IPP,IPSS,VPSS

INTERVENTIONS:
Diagnostic Test: IPP,IPSS,VPSS — Prostate volume, IPSS, VPSS and IPP were determined after urological examinations of the patients.

SUMMARY:
The diagnosis of bladder outlet obstruction is made by pressure-flow studies, which is an invasive method. This study was conducted to evaluate non-invasive, effective, and low-cost diagnostic methods in male patients with bladder filling and emptying abnormalities.

DETAILED DESCRIPTION:
Aims The diagnosis of bladder outlet obstruction is made by pressure-flow studies, which is an invasive method. This study was conducted to evaluate non-invasive, effective, and low-cost diagnostic methods in male patients with bladder filling and emptying abnormalities.

Methods The study included 219 male patients aged 50 and over, who were admitted between March 2020 and August 2020. Patients completed the Visual Prostate Symptom Score (VPSS) along with International Prostate Symptom Score (IPSS). Intravesical prostatic protrusion (IPP), prostate volume, bladder volume, and post voiding residual urine (PVR) were measured by suprapubic ultrasound. Urethral resistance was calculated using the Bladder Outlet Obstruction Number (BOON), and patients over -20 were considered obstructed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of BPH Disease

Exclusion Criteria:

* Patients with previous urological surgery
* History of urological malignancy
* Systemic disease (diabetes mellitus, multiple sclerosis, etc.)
* Trauma that may cause LUTS
* Pharmacotherapy for LUTS
* Use diuretic antihypertensive
* PSA > 4 ng/dl
* History of pelvic radiotherapy
* Visual problems that could not complete the VPSS test were not included.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Male patients over 50 years old who applied to Sivas Cumhuriyet University Hospital urology outpatient clinic between March 2020 and August 2020.
Sampling Method: Non-Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
The Importance of Non-invasive Methods in the Diagnosis of Lower Urinary System Symptoms. | During the patient's outpatient clinic examination
  In this study, it is aimed to determine the use of VPSS instead of IPSS when needed, the importance of IPP in evaluating LUTS, and the correlation of IPP with VPSS and IPSS, based on BOON in the diagnosis of obstruction.
  The data obtained from the study were evaluated with the SPSS 23.0 program. The normality rankings of the data were made by the Shapiro-Wilk test. Since the data are non-parametric, the Spearman correlation test was performed. The Kruskal-Wallis test was performed for calculating the difference of IPSS groups (mild, moderate, severe) according to other parameters. In case of difference, the Mann-Whitney U test was applied to understand which two groups were different. Since the IPP groups (<5mm, 5-10mm, >10mm) conformed to the normal distribution, Post-Hoc (Bonferroni) test was used to determine the differences between the 3 groups. The level of error was taken as 0.05.

CONTACTS AND LOCATIONS:
Locations (1):
- Cumhuriyet Universty, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code